CLINICAL TRIAL: NCT04002271
Title: Acute Postoperative Pain Control After Robotic Arm Assisted Total Knee Replacement: a Randomized Controlled Trial Comparing Three Anaesthetic Techniques
Brief Title: Total Knee Replacement TIVA With Robotic Arm Assisted
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW19-282
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain
Keywords: TIVA; total knee replacement; post operative pain; acute pain; anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Propofol; Sevoflurane; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Patients in group SA will undergo spinal anaesthesia. Patients in group GAS will undergo general inhalational anaesthesia using sevoflurane. Patients in group TIVA will undergo general anaesthesia using propofol total intravenous anaesthesia
Who Masked: Investigator
Masking Description: This is an observer blinded randomized controlled trial. The patients will be aware of whether they received spinal anaesthesia (SA) or general anaesthesia (TIVA or GAS). The investigators responsible for assessing outcomes and collecting data will be blinded to patient allocation. The anaesthetist performing anaesthesia will be aware of patient allocation, but will not be involved in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group SA (Active Comparator): Patients in Group SA will undergo spinal anaesthesia.
  Interventions: Procedure: Spinal anaesthesia
- Group GAS (Active Comparator): Patients in Group GAS will undergo general inhalational anaesthesia using sevoflurane.
  Interventions: Drug: Sevoflurane
- Group TIVA (Experimental): Patients in Group TIVA will undergo general anaesthesia using propofol total intravenous anaesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Target controlled infusion (TCI) with modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia. Level of anaesthesia will be titrated to produce a BIS value of between 40-60. For induction, remifentanil 1mcg/kg and rocuronium 0.6 mg/kg will be given intravenously prior to intubation. Sevoflurane will not be given. Air and oxygen will be given, and FiO2 will be kept at between 35-50%. Similarly, to the GAS group, remifentanil will be infused at a rate of between 0.1-0.2mcg/kg/min and titrated according to the haemodynamic parameters stated for the GAS group. Morphine sulphate will be given at a dose of 0.1mg/kg before skin incision. TCI propofol and remifentanil will be switched off at the end of the procedure. Reversal of muscle relaxation will be achieved as for the GAS group.
  Arms: Group TIVA
Drug: Sevoflurane — Patients in the GAS group will be induced with intravenous bolus propofol 1.5-3mg/kg, remifentanil 1mcg/kg, and rocuronium 0.6mg/kg for induction of general anaesthesia and intubation of patient. General anesthesia monitoring will be used. Maintenance of general anesthesia to be provided using sevoflurane, together with air and oxygen. FiO2 will be maintained between 35-50%. Bispectral (BIS) monitoring will be applied and level of anaesthesia will be maintained at a BIS value of 40-60. Remifentanil infusion will be given at between 0.1-0.2mcg/kg/min, to be titrated to maintain mean arterial blood pressure within 20% of baseline (blood pressure in ward before surgery as baseline) and heart rate between 45 to 100 bpm. Morphine sulphate to be given at a dose of 0.1mg/kg before skin incision. Sevoflurane and remifentanil infusion will be switched off at the end. Reversal of muscle relaxation to be achieved using intravenous neostigmine 50mcg/kg and atropine 20mcg/kg after the operation.
  Arms: Group GAS
Procedure: Spinal anaesthesia — Patients in the SA group will receive intrathecal (L4-5, or L3-4 if failed at L4-5) administration of 2.2-2.4ml 0.5% heavy bupivicaine using a 25G Whitacare needle. No intrathecal opioid will be given during the procedure. Light sedation will be given during surgery with target-controlled infusion of propofol using the Marsh effect site model (0.3 -1 mcg/ml). Supplemental oxygen 2L/min will be given via the nasal cannula.
  Arms: Group SA

SUMMARY:
Total knee replacement (TKR) is a commonly performed surgical procedure, and is associated with moderate to severe acute postoperative pain. Poor acute postoperative pain control has been associated with increased morbidity, prolonged recovery, reduced patient satisfaction and chronic post-surgical pain. Multimodal analgesia in the context of enhanced recovery after surgery programs is advocated for conventional total knee replacement. More recently, robotic arm assisted total knee replacement has been introduced. TKR is most commonly performed under spinal anaesthesia or general anaesthesia using inhalational agents or propofol total intravenous anaesthesia (TIVA). It is unclear which is the best anaesthetic technique for postoperative analgesia. There has been no head to head trial comparing these 3 anaesthetic techniques in the context of modern multimodal and enhanced recovery after surgery (ERAS) protocols for conventional and robotic arm assisted TKR. Propofol TIVA may reduce postoperative pain and opioid consumption after surgery, but the overall evidence is still controversial. Whether propofol TIVA provides better analgesia compared to inhalational anaesthesia for TKR is not known. A prospective, randomized controlled trial providing head to head comparisons between general anaesthesia with propofol TIVA, inhalational anaesthesia, and spinal anaesthesia under is indicated.

In this study, we plan to perform a randomized controlled trial to compare postoperative analgesia after robotic arm assisted TKR in three commonly used anaesthetic techniques: 1) spinal anaesthesia (SA), 2) general anaesthesia with inhalational anaesthesia (GAS), 3) general anaesthesia with propofol TIVA (TIVA). This clinical trial will be conducted within the framework of modern multimodal analgesic and enhanced recovery after surgery pathways.

In this study, we plan to perform a randomized controlled trial to compare postoperative analgesia after TKR in three commonly used anaesthetic techniques: 1) spinal anaesthesia (SA), 2) general anaesthesia with inhalational anaesthesia (GAS), 3) general anaesthesia with propofol TIVA (TIVA). This clinical trial will be conducted within the framework of modern multimodal analgesic and enhanced recovery after surgery pathways.

DETAILED DESCRIPTION:
Preoperative Care

Patients will be approached at the preadmission clinic or in the general ward before operation. The anaesthetic techniques will be explained and s/he will be recruited into the study if s/he agrees. Fasting will start 6 hours before surgery for solids and 2 hours clear fluid. All patients will be given oral celebrex 200mg, paracetamol 1g and pregabalin 50mg po, two hours before start of anaesthesia.

Range of movement of the operating knee, quadriceps function, pain scores of the affecting knee will be assessed on day before operation. Baseline data for health related quality of life, psychological status, and quality of recovery will be obtained using the Chinese Hong Kong version of SF-36, Depression Anxiety Stress Scales (DASS) and the Chinese quality of recovery (QoR) score, respectively.

Anaesthesia and intraoperative care

On arrival to the operation theatre, a 18 or 16 gauge intravenous cannula will be inserted. Standard monitoring with pulse oximeter, non-invasive blood pressure, and three lead electrocardiogram will be applied before start of anaesthesia. Non-invasive blood pressure will be checked at least every 5 minutes throughout the operation.

Spinal anaesthesia (SA) group

Patients in the SA group will receive intrathecal (L4-5, or L3-4 if failed at L4-5) administration of 2.2-2.4ml 0.5% heavy bupivicaine using a 25G Whitacare needle. No intrathecal opioid will be given during the procedure. Light sedation will be given during surgery with target-controlled infusion of propofol using the Marsh effect site model (0.3 -1 mcg/ml). Supplemental oxygen 2L/min will be given via the nasal cannula.

General anaesthesia with inhalational anaesthesia (GAS) group

Patients receiving inhalational general anaesthesia will be induced with intravenous bolus propofol 1.5-3mg/kg, remifentanil 1mcg/kg, and rocuronium 0.6mg/kg for induction of general anaesthesia and intubation of the patient. General anesthesia monitoring will be used. Maintenance of general anesthesia would be provided using sevoflurane, together with air and oxygen. FiO2 will be maintained between 35-50%. Bispectral (BIS) monitoring will be applied and level of anaesthesia will be maintained at a BIS value of between 40-60. Remifentanil infusion will be given at between 0.1-0.2mcg/kg/min. This will be titrated to maintain mean arterial blood pressure within 20% of baseline (blood pressure in the ward before surgery will be taken as baseline) and heart rate between 45 to 100 beats per minute. Muscle relaxants can be given as required. Morphine sulphate will be given at a dose of 0.1mg/kg before skin incision. Sevoflurane and remifentanil infusion will be switched off at the end of the procedure. Reversal of muscle relaxation will be achieved using intravenous neostigmine 50mcg/kg and atropine 20mcg/kg after the operation.

General anaesthesia with propofol total intravenous anaesthesia (TIVA) group

Target controlled infusion (TCI) with modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia. Level of anaesthesia will be titrated to produce a BIS value of between 40-60. For induction, remifentanil 1mcg/kg and rocuronium 0.6 mg/kg will be given intravenously prior to intubation. Sevoflurane will not be given. Air and oxygen will be given, and FiO2 will be kept at between 35-50%. Similarly, to the GAS group, remifentanil will be infused at a rate of between 0.1-0.2mcg/kg/min and titrated according to the haemodynamic parameters stated for the GAS group. Morphine sulphate will be given at a dose of 0.1mg/kg before skin incision. TCI propofol and remifentanil will be switched off at the end of the procedure. Reversal of muscle relaxation will be achieved as for the GAS group.

Intraoperative care for all 3 groups

Intravenous antibiotic will be given before skin incision. Hypotension will be managed with intravenous phenylephrine or ephedrine at the discretion of the anaesthesiologist. Hypertension or tachycardia in patients from the TIVA and GAS groups will be managed by titrating the remifentanil infusion up to 0.2mcg/kg. Intravenous anti-hypertensive drugs such as beta-blockers (eg esmolol, metoprolol), hydralazine, glyceryl trinitrate and phentolamine can be given if hypertension persists. Intra-operative fluid 8-10ml/kg/hr will be infused as maintenance. In addition, fluid replacement will be given for of blood loss. Infusion fluid warmer and thermal blankets will be used with the aim of keeping a core temperature of 35.5-37.5 degrees Celsius. All patients will be given 4mg of intravenous ondansetron 30 minutes before end of surgery.

Local anaesthetic infiltration with 40ml 0.75% ropivacaine, 0.5ml 1:200,000 adrenaline, 30mg ketorolac in 60ml normal saline over the perisurgical area will be administrated by orthopaedic surgeon after implant insertion and wound closure.

Patients will subsequently be transferred to the post anaesthetic care unit (PACU) for monitoring for at least 1 hour.

Analgesic modalities and assessment

Procedures for all the analgesic modalities are described below:

For all the groups

Resting numerical rating scale (NRS) pain scores will be checked every 5 minutes in the PACU. In the PACU, 2mg intravenous morphine will be given every 5 minutes until the numerical rating pain score (NRS) is less than 4/10. Patient controlled analgesia (PCA) with morphine will then be given once NRS is less than 4/10. The PCA device will be configured to give 1 mg of bolus dose of morphine with each demand and the lockout duration will be 5 minutes. No background infusion will be given and the maximum dose limit of morphine will be 0.1mg/kg per hour. Intramuscular morphine sulphate at a dose of 0.1mg/kg will be prescribed every 4 hours if necessary, for breakthrough beginning from postoperative day (POD) 0. Intravenous 4mg ondansetron every 4 hours as necessary will be prescribed for nausea or/and vomiting. While in the PACU, the respiratory rate, oxygen saturation, Ramsay sedation scores, blood pressure and heart rate will be monitored every 5 minutes.

On POD 0, patients will resume oral diet if not contraindicated. Oral paracetamol 1g tds, celebrex 200mg daily, and pregabalin 50mg once at night will be given to all patients for 5 days. Dihydrocodeine 30mg q6h po prn for 5 days will be prescribed after cessation of PCA morphine.

While on PCA morphine, the patient's respiratory rate, SpO2 and sedation score will be monitored every hour. Heart rate and blood pressure will be checked every 4 hours. NRS pain scores at rest, during knee movement (knee flexion), cumulative PCA morphine doses, and number of PCA demands/goods delivered, and side effects (eg nausea, vomiting, dizziness, pruritis) will be recorded every 4 hours. Patients will be assessed by the pain team every day.

Patients will be on PCA morphine for 2 days. If NRS pain scores during knee movement on POD 2 is less than 4/10 and morphine consumption is low, PCA morphine will be stopped. PCA morphine will be continued if NRS pain score is equal or greater than 4, or if PCA morphine consumption is high. After cessation of PCA morphine, NRS pain scores at rest and during knee movement, as well as the dose and frequency of rescue analgesia and the incidence of side effects will be charted once a day until discharge. Patient satisfaction with analgesia (0-10, where 0 is the least satisfaction, and 10 is the most satisfaction) will be assessed daily during hospital stay. Overall benefit of analgesic scores (OBAS) will be checked once a day.

Phone follow up will be done for all patients on POD 3, 4, and 5 (if patient discharged home on those days). NRS pain scores at rest and with movement, analgesic medication consumption (pill count), incidence of adverse side effects (nausea, vomiting, pruritis, dizziness), and OBAS.

Surgical technique/Prosthesis

The surgery will be performed by the same surgical team with standardized surgical technique. All the patients will have posterior stabilized knee prosthesis. Tranexamic acid will be given according to protocol. Standardized regimen and technique of local infiltration of analgesic at the end of the surgery will be given as part of the multi-modal pain control protocol.

Postoperative care and assessment

POD 0 mobilization or early mobilization with physiotherapy and occupational therapy rehabilitation is encouraged after operation. Fluid diet will be allowed on POD 0. The surgical team will assess for occurrences of postoperative surgical complications, suitability for discharge (good pain control, ambulation, normal bowel function, and ability to eat properly without vomiting. Urinary retention will be documented as well. Time to mobilization and time to soft diet intake will be recorded. Active and passive range of movement of the operated knee, ability to achieve straight leg raising, and other rehabilitation parameters will be assessment by allied health staffs from POD 0 till day of discharge. Sleep disturbance due to pain (0-10, where 0 represents no disturbance and 10 represents the most disturbance possible) and quality of recovery (Chinese QoR) will be assessed on POD 1 and 2.

Postoperative follow up (3 months, 6 months)

Questions about pain that will be asked during the face-to-face interview at 3 months, 6 months. Chronic post-surgical pain will be assessed based on the core outcome set recommended by Wylde et al, which is specific for total knee replacement:

* The presence or absence of chronic pain (yes/no)
* Pain intensity (NRS pain score, 0-10): at rest, during movement of the ipsilateral knee
* Pain and physical functioning: pain with general activity, with walking, when kneeling, climbing stairs, descending stairs (NRS 0-10)
* Temporal aspects of pain: frequency breakthrough pain (NRS pain score over 6/10), duration of pain since operation, night pain, constant pain.
* Pain description: location of the pain: medial or lateral aspect of knee, scar; pain quality
* Identification Pain Questionnaire to test for neuropathic pain
* Any analgesic consumption: yes/no, frequency of use (eg number of times analgesics taken per week), type of medication used, dose of medication used.
* Patient Global Impression of Change Scale (PGIC)
* Health related quality of life (Chinese SF-36)
* Depression Anxiety Stress Scale (DASS)
* Pain self-efficacy questionnaire
* Effect of pain on sleep disturbance (0-10)

Physical examination

* Range of motion of the knee
* Any area of decreased sensation, brush allodynia and pinprick hyperalgesia at the ipsilateral knee, scar site.
* KSKS and KSK functional score (done by physiotherapist and occupational therapist)

Blood taking

Blood taking will be performed to check for the levels of potential pain mediators. These include PTEN, TNF-α, IL-6, and IL-β. These will be collected just before surgery (during induction of anaesthesia), on POD 0 and POD1.

Other Data collection

The following data will be collected during the perioperative period:

* Demographics
* Time of admission
* Intraoperative vital signs (blood pressure, heart rate, oxygen saturation)
* Estimated intraoperative blood loss
* Tourniquet time if any
* Volume of intraoperative fluid/blood infusion
* Duration of surgery and anaesthesia
* Time of discharge

If at certain time point after operation, the patients cannot be managed according to the protocol due to any reason such as the development of complication, no further data will be collected. These patients will still be followed up. Intention-to-treat analysis will be used. Patients will remain in their initial designated groups for data analysis even if there is a change in surgical or anaesthetic/analgesic management, as long as they have had unilateral total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Scheduled for elective primary unilateral total knee replacement
* Able to speak and understand Chinese (including Cantonese and Mandarin)
* Able to provide informed consent

Exclusion Criteria:

* Revision total knee replacement
* Single stage bilateral total knee replacement
* Previous major knee surgery to the same knee
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* Rheumatoid arthritis
* Immunological depression
* Chronic opioid user
* Alcohol or drug abuse
* Obesity (Body mass index over 35kg/m2)
* Impaired liver function (Plasma bilirubin over 34 μmol/L, INR ≥ 1.7, ALT and AST over 100U/L)
* Impaired renal function, defined as preoperative serum creatinine level over 120 μmol/L
* Pre-existing neurological or muscular disorders
* Psychiatric or neurological disease that could potentially influencing pain perception
* Impaired or retarded mental state
* Difficulties in using patient controlled analgesia (PCA)
* Pregnancy
* Local infection
* Patient refusal
* Strong preference for a particular type of anaesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by numerical rating scales (NRS) pain scores | from postoperative day 0 until postoperative day 4
  NRS pain scores (from 0-10, where 0 is the least satisfaction and 10 most satisfaction) will be recorded at rest and with movement everyday.

SECONDARY OUTCOMES:
PCA morphine consumption | from postoperative day 0 until postoperative day 5
  Cumulative PCA morphine doses (in mg) will be recorded daily based on medical record.
Dihydrocodeine use | from postoperative day 0 until postoperative day 5
  Frequency of dihydrocodeine use (i.e. how many times per day) will be recorded daily
Side effects of analgesics | from postoperative day 0 until postoperative day 5
  Pruritus, dizziness, nausea, vomiting, wound infection, urinary retention, confusion
Range of motion (ROM) of knee | until postoperative day 6
  Active and Passive ROM of knee (flexion and extension) will be recorded.
Overall benefit of analgesic scores (OBAS) | from postoperative day 0 to postoperative day 5 on phone
Effect of pain on sleep disturbance | from postoperative day 1 to postoperative day 2, follow-up in 3 months, 6 months
  (0-10, where 0 represents no disturbance and 10 represents the most disturbance possible

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong